CLINICAL TRIAL: NCT01758939
Title: Phase 4 Predictors of Response to Combined Pegylated Interferon and Ribavirin in Chronic Hepatitis C Genotype IV Infected Egyptian Patients
Brief Title: Predictors of Response to Combined Pegylated Interferon and Ribavirin in Chronic Hepatitis C Infected Egyptian Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Zekri AR, Proffesor, Cairo University
Other Study IDs: 2; NZEKRI2 (Registry Identifier: NZEKRI)
Record Dates: First submitted 2012-12-25; First posted 2013-01-01 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Hepatitis C, Chronic
Keywords: Peg Interferon,; Ribavirin,; HCV,; Genotype IV.
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hepatitis C virus infected patients

SUMMARY:
Retrospective prospective cohort study aimed at Assessing the predictors to the response to the antiviral combined therapy with pegylated Interferon (Both types: Alfa 2 A and Alfa 2 B) in hepatitis C virus infected Egyptian patients.

DETAILED DESCRIPTION:
Retrospective prospective cohort study conducted on HCV infected patients treated with Interferon alpha therapy, the retrospective part of the study includes the data of the patients retrieved from medical records from the period from September 2006 till January 2011. Then from January 2011 the study became prospective national study. Responders to therapy were defined by normalization of serum alanine aminotransferase (ALT) and absence of detectable serum HCV RNA at the end of treatment (48 weeks). Relapsed responders to therapy were defined by normalization of serum ALT and absence of detectable serum HCV RNA at the end of treatment but with an increase of the serum ALT and the presence of HCV RNA at follow-up 72 weeks). Non-responders were defined by elevated serum ALT and the presence of HCV RNA at the end of treatment. All patients will sign a written informed consent to share in this clinical registry by their data and biological samples. Sub-studies will be conducted on subgroups of patients sharing in this main study after signing a written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Age: above eighteen years and below 60

  * Detectable HCV RNA in serum by PCR
  * ALT level ranged from normal to three fold elevation.
  * Minimum hematological values of hemoglobin of 10.5 g/dl for females, 12g/dl for males; white blood count 3×109/L; platelet counts not less than 100,000/mm3.
  * Bilirubin, albumin, prothrombin time and creatinine within normal limits.
  * A suitable method for assessment of fibrosis lik liver biopsy or fibroscan will be done before the start of treatment to assess the degree of necroinflammatory response to HCV, which was further subgrouped by HAI scoring system into mild, moderate & severe.

Exclusion Criteria:

* Decompensated cirrhosis
* Other causes of liver diseases
* Autoimmune disorders
* Uncontrolled diabetes
* Thyroid dysfunction
* Neurological or cardiovascular disease
* Malignancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: chronic hepatitis C virus , genotype IV, infected Egyptian patients
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2011-01; Primary Completion 2016-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Assess the response to the Interferon therapy. | After 72 weeks of the start of therapy of each patient

SECONDARY OUTCOMES:
Predictors of response to therapy | at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Gamal Esmat, MD, Principal Investigator — Cairo University; Abdelrahman Zerki, PHD, Principal Investigator — Cairo University; Wahid Doss, MD, Study Director — Cairo University; Maissa El Raziky, MD, Study Chair — Cairo University; Gamal Sheha, MD, Study Chair — Cairo University; Tarneem Darwish, MSc., Study Chair — Cairo University; samy zaki, MD, Study Chair — Cairo University; Magdi El-Serafy, MD, Study Chair — Cairo Universty; Fathalla Sedky, MD, Study Chair — Cairo University; Ahmed M Nasr, MD, Study Chair — Cairo University; Mostafa Gabr, MD, Study Chair — Cairo University; Ali kassem, MD, Study Chair — Cairo University; Ibrahim Metawea, MD, Study Chair — Cairo University; Noaman Al-Garem, MD, Study Chair — Cairo University; Hassan Hamdy, MD, Study Chair — Cairo University; Tawheed Mwafy, MD, Study Chair — Cairo University; Khalil A Khalil, MD, Study Chair — Cairo University; Magdy Atta, MD, Study Chair — Cairo University; Osama E Salem, MD, Study Chair — Cairo University; Mohamed A Afify, MD, Study Chair — Cairo University; Mohamed S Al-Shazly, MD, Study Chair — Cairo University; Hamdy Mahfouz, MD, Study Chair — Cairo University; Mustafa Gabr, MD, Study Chair — Cairo University; Monquez Motaea, MD, Study Chair — Cairo University; Hossam Abdel-Latif, MD, Study Chair — Cairo University
Locations (1):
- Viral Hepatitis Treatment Units affiliated to National Committee for Control of Viral Hepatitis, Cairo, Cairo Governorate, Egypt

REFERENCES:
- [Derived] N Zekri AR, Raafat AM, Elmasry S, Bahnassy AA, Saad Y, Dabaon HA, El-Kassas M, Shousha HI, Nassar AA, El-Dosouky MA, Hussein N. Promotor methylation: does it affect response to therapy in chronic hepatitis C (G4) or fibrosis? Ann Hepatol. 2014 Sep-Oct;13(5):518-24. PMID 25152984
- [Derived] Zekri AR, Bahnassy AA, Mohamed WS, Alam El-Din HM, Shousha HI, Zayed N, Eldahshan DH, Abdel-Aziz AO. Dynamic interplay between CXCL levels in chronic hepatitis C patients treated by interferon. Virol J. 2013 Jul 1;10:218. doi: 10.1186/1743-422X-10-218. PMID 23816271